CLINICAL TRIAL: NCT02889835
Title: "Clinical Performance of an Incrementally Placed Highly Filled Composite, an Incrementally Placed Flowable Composite, and a Bulk Filled Composite in Class II Restorations"
Brief Title: Clinical Performance of Incremental and Bulk Fill Composites in Class II Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CR16-005
Record Dates: First submitted 2016-04-27; First posted 2016-09-07 (Estimated); Results first posted 2023-09-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
Keywords: Class II; molar and premolar; resin composite; adult; restoration
MeSH Terms: conditions — Dental Caries; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Intervention Model Description: Single group with a split mouth design in which each subject received all three treatments. Of the 53 total subjects, 3 study subjects actually received duplicate treatment, i.e., they received 6 dental restorations.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Universal Composite (Active Comparator): Supreme Universal Restorative
  Interventions: Device: Supreme Universal Restorative
- Flowable Composite (Experimental): Supreme Flowable Restorative
  Interventions: Device: Supreme Flowable Restorative
- Bulk Fill Flowable Composite (Experimental): Bulk Fill Flowable Restorative
  Interventions: Device: Bulk Fill Flowable Restorative

INTERVENTIONS:
Device: Supreme Universal Restorative
  Arms: Universal Composite
Device: Supreme Flowable Restorative
  Arms: Flowable Composite
Device: Bulk Fill Flowable Restorative
  Arms: Bulk Fill Flowable Composite

SUMMARY:
This study will examine the clinical performance of Class II restorations over a three year period with 3 composite resins - a conventional composite resin, a flowable composite resin and a bulk placed and cured composite resin.

DETAILED DESCRIPTION:
Specific Aim: To place three commercially available resin composites in Class II cavity preparations of adult patients, evaluate the resin composite restorations at baseline, 6 months, 1 year, 2 and 3 years using specific criteria defined by International Dental Federation (FDI).

ELIGIBILITY:
Inclusion Criteria:

* must have given written informed consent to participate in the trial
* must need at least three posterior dental fillings
* replacement restorations due to caries or an esthetic replacement with or without caries are acceptable.
* must be available for the required post-operative follow-up visits
* restorations must be in contact with opposing natural or crowned teeth with at least at least one occlusal contact in habitual closure
* Class II restorations must have at least one proximal contact
* restorations must have a buccal to lingual/palatal width no greater than 1/3 the distance from buccal to lingual/palatal cusp tips
* all restorations must Class II with a proximal contact with a natural or artificial tooth

Exclusion Criteria:

* have severe medical complications (organ transplants, long term antibiotic or steroid treatment, cancer or immunocompromised) and disabilities who may not be able to tolerate the time required to complete the restorations or to provide adequate oral hygiene
* have xerostomia either by taking medications known to produce xerostomia or those with radiation induced or Sjogren's syndrome patients
* have chronic periodontitis, rampant caries or poor oral hygiene which may require extraction of the teeth to be restored
* are unavailable for long term recall
* cannot tolerate the rubber dam required for isolation of the tooth during preparation and restoration.
* do not meet all inclusion criteria
* present with any systemic or local disorders that contra-indicate the dental procedures included in this study
* have an unstable occlusion
* have severe bruxing or clenching or in need of TMJ related therapy
* have teeth with periapical pathology or expected pulp exposures
* have teeth that are non-vital or that exhibit signs of pulpal pathology
* are pregnant.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Lawson, DDS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Dental School, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 53 subjects were evaluated at baseline (3 subjects with 2 sets of restorations). "Number Started" will be greater than the Protocol Enrollment and cannot be revised, however, this is acceptable for split-person studies.
Units Other Than Participants: Teeth
Groups:
- Universal Composite; Flowable Composite; Bulk-fill Composite: This is a split-mouth design with each subject receiving one or two replicates of each of three restorative dental-filling materials: 1) Supreme Universal Composite, 2) Supreme Flowable Composite, and/or, 3) Bulk-fill Composite
Period: Overall Study
Arm/Group | Universal Composite | Flowable Composite | Bulk-fill Composite
Started (A total of 53 patients were enrolled. Each patient received in different teeth, one restoration of each intervention except for 3 patients who received two restorations of each intervention for a total of 56 teeth per intervention.) | 53; 56 Teeth | 53; 56 Teeth | 53; 56 Teeth
Completed | 35; 37 Teeth | 35; 37 Teeth | 35; 37 Teeth
Not Completed | 18; 19 Teeth | 18; 19 Teeth | 18; 19 Teeth
Not completed — Lost to Follow-up | 13 | 13 | 13
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Exclusion Criteria -change in oral status | 1 | 1 | 1
Not completed — Death | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: A total of 53 patients were enrolled. Each patient received in different teeth, one restoration of each intervention except for 3 patients who received two restorations of each intervention for a total of 56 teeth per intervention.
Units Other Than Participants: Teeth
Groups:
- Universal Composite, Flowable Composite, Bulk Fill Flowable Composite: Split-mouth design where each enrolled subject received one or two replicates of three restorative materials: 1) Supreme Universal Restorative, 2) Supreme Flowable Restorative, and/or, 3) Bulk Fill Flowable Restorative
Arm/Group | Universal Composite, Flowable Composite, Bulk Fill Flowable Composite
Number analyzed (Participants) | 53
Number analyzed (Teeth) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Percent Acceptable Restorations
Description: Percentage of restorations that survived (percent clinically acceptable per FDI criteria) over 36 months.
Time Frame: 36 Months
Measure: Number; unit: percentage of restorations survived
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 53 | 54 | 52
Number analyzed (Teeth) | 53 | 54 | 52
percentage of restorations survived | 94.6 | 96.4 | 92.9
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Kaplan-Meier analysis was performed to assess survival over 36 months. Test of survival distributions for the three arms were calculated using Log Rank (Mantel-Cox). Sample size is based on guidelines of the American Dental Association for obtaining approval as an amalgam replacement for posterior restorations - minimum of 40 restorations in a minimum of 20 subjects at 18 months. Sample size is based by taking subject attrition into account over the 36 month clinical evaluation; Test type: Superiority; p = 0.686, Log Rank

2. Secondary Outcome: Surface Luster
Description: 1. Luster comparable to enamel
  2. Slightly dull, not noticeable from speaking distance.
  3. Surface is dull but still acceptable if the surface of the restoration is covered with a film of saliva.
  4. Surface is rough and not masked by salivary film. Major re-finishing or veneering is necessary and possible.
  5. Surface is unacceptably rough which makes it ugly and/or it retains noticeable biofilm (plaque). Improvement by finishing or veneering is not feasible.
Time Frame: 36 Month
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.50 (0.58) | 1.39 (0.57) | 1.41 (0.50)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.701, Kruskal-Wallis

3. Secondary Outcome: Surface Staining
Description: 1. No surface staining.
  2. Minor surface staining (under dry conditions) is present but is evenly spread over all the teeth. It does not affect the aesthetic properties because it is generalized and acceptable.
  3. Moderate surface staining not noticeable from a speaking distance.
  4. Surface staining is present on the restoration but not the tooth and is clearly recognizable from a speaking distance. The aesthetic properties of the dentition are affected. Restoration requires major correction and layering of new material.
  5. Surface staining is totally unacceptable/unsightly and the restoration needs to be replaced.
Time Frame: 36 Month
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.21 (0.50) | 1.25 (0.44) | 1.19 (0.40)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.812, Kruskal-Wallis

4. Secondary Outcome: Color Match
Description: 1. Colour and translucency of the restoration have a clinically excellent match with the surrounding enamel and adjacent teeth. There is no difference in shade, brightness or translucency between restoration and tooth.
  2. Colour match is clinically acceptable but minor deviations in shade between tooth and restoration are apparent.
  3. Colour match is satisfactory; there is a clear deviation in colour match that does not affect aesthetics.
  4. Colour match is satisfactory; there is a clear deviation in colour match that does not affect aesthetics.
  5. Colour match and/or translucency are clinically unsatisfactory. The restoration displays an unacceptable alteration in colour and/or translucency. Restoration needs replacement.
Time Frame: 36 Month
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.36 (0.49) | 1.32 (0.48) | 1.67 (0.73)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.104, Kruskal-Wallis

5. Secondary Outcome: Fracture of Material and Retention
Description: 1. No fractures / cracks.
  2. Small hairline crack.
  3. Two or more or larger hairline cracks and/or material chip fracture not affecting the marginal integrity or approximal contact.
  4. Material chip fractures which damage marginal quality or approximal contacts.
  5. Bulk fractures with partial loss (less than half of the restoration).
Time Frame: 36 Month
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.21 (0.79) | 1.07 (0.38) | 1.04 (0.19)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.440, Kruskal-Wallis

6. Secondary Outcome: Occlusal Wear - Qualitative
Description: 1. Physiological wear equivalent to enamel.
  2. Normal wear only slightly different from that of enamel.
  3. Different wear rate than enamel but within the biological variation.
  4. Wear considerably exceeds normal enamel wear; or occlusal contact points are lost.
  5. Wear considerably exceeds normal enamel wear; or occlusal contact points are lost.
Time Frame: 36 Month
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.14 (0.36) | 1.07 (0.26) | 1.11 (0.32)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.676, Kruskal-Wallis

7. Secondary Outcome: Tooth Integrity
Description: 1. Complete integrity.
  2. Small marginal enamel fracture (<150 µm) / Hairline crack in enamel (<150 µm)
  3. Marginal enamel defect <250µm / Crack <250µm / Enamel chipping
  4. Multiple cracks / Major marginal enamel defects; gap > 250 µm or dentine or base exposed
  5. Cusp or tooth fracture
Time Frame: 36 Month
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.00 (0) | 1.00 (0) | 1.00 (0)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 1.000, Kruskal-Wallis

8. Secondary Outcome: Recurrence of Caries, Erosion, Abfraction
Description: 1. No secondary or primary caries
  2. Small and localized: Demineralization / Erosion / Abfraction.
  3. Larger areas of: Demineralisation / Erosion / Abrasion / abfraction, dentine not exposed. Only preventive measures necessary
  4. Caries with cavitation and suspected undermining caries / Erosion in dentine / Abrasion, abfraction in dentine. Localized and accessible can be repaired.
  5. Deep caries or exposed dentine that is not accessible for repair of restoration
Time Frame: 36 Months
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.15 (0.60) | 1.11 (0.57) | 1.04 (0.19)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.764, Kruskal-Wallis

9. Secondary Outcome: Margin Adaptation
Description: 1. No clinically detectable gap.
  2. Marginal integrity deviates from ideal but could be upgraded to ideal by polishing.
  3. Leakage/discoloration is present but limited to border area of margins. Generalized marginal gap >150 µm but <250 µm, easily perceptible on probing but cannot be modified without minor damage to tooth or surrounding tissue, and is not considered to result in long-term negative consequences for tooth or surrounding tissue if left untreated. Presence of several small marginal fractures that are unlikely to cause long-term effects.
  4. Localized gap larger than 250 µm, may result in exposure of dentine or base. Repair necessary for prophylactic reasons.
  5. Generalized gap larger than 250 µm or restoration is loose but in situ, replacement necessary or large fractures at margins and loss of material is too extensive to be repaired.
Time Frame: 36 Months
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.41 (0.57) | 1.21 (0.42) | 1.33 (0.55)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.323, Kruskal-Wallis

10. Secondary Outcome: Marginal Staining
Description: 1. No marginal staining
  2. Minor marginal staining, easily removable.
  3. Moderate marginal staining, not aesthetically unacceptable.
  4. Pronounced (mainly localized) marginal staining and not removable by polishing; major intervention necessary for improvement. of aesthetics
  5. Deep marginal staining (generalized and/or profound), not accessible for intervention.
Time Frame: 36 Months
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.33 (0.59) | 1.29 (0.53) | 1.26 (0.59)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.714, Kruskal-Wallis

11. Secondary Outcome: Proximal Contact Point
Description: 1. Contact is physiological (dental floss can only be inserted into the interdental space under pressure).
  2. Contact is slightly too strong but acceptable. Floss or 25 µm metal blade can only be passed through contact with force/pressure.
  3. Contact is weak, a 50 µm metal blade can pass through contact area but not a 100 µm blade, or floss passes very easily with only a slight snap effect. There is no indication for removing/repairing restoration and there is no damage to tooth, gingiva or other periodontal structures. There is no cervical caries, inflammation of the gingival papilla through food impaction, or pocket formation.
  4. Contact is weak and a 100 µm metal blade can easily pass through. In addition there are signs of damage to tooth (i.e. cervical caries,). Repair is necessary.
  5. Contact is weak allowing damage due to food impaction and demonstrating pain/gingivitis requires immediate intervention. Repair is not feasible and replacement is necessary.
Time Frame: 36 Months
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.17 (0.58) | 1.17 (0.58) | 1.10 (0.45)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.846, Kruskal-Wallis

12. Secondary Outcome: Patient's View
Description: 1. Entirely satisfied with aesthetics and function
  2. Satisfied with aesthetics and function
  3. Minor criticism but no adverse clinical effects.
  4. Desire for improvement (aesthetics / function); Reshaping of anatomic form or refurbishing is possible.
  5. Completely dissatisfied and / or adverse effects, incl. pain
Time Frame: 36 Months
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.0 (0.00) | 1.0 (0.00) | 1.0 (0.00)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 1.000, Kruskal-Wallis

13. Secondary Outcome: Post-op Sensitivity
Description: 1. No postoperative hypersensitivity. Normal pulp vitality response.
  2. Postoperative hypersensitivity of short duration (less than one week) and no longer present at the baseline assessment. Pulp vitality response normal at baseline assessment (one week after placement).
  3. Intense postoperative hypersensitivity of duration greater than one week but less than six-months.
  4. Persistent postoperative hypersensitivity. Response to cold stimulus is markedly premature/strong and major intervention is necessary; or there is extremely delayed/weak and unclear or negative sensitivity. Sensitivity level is significantly different from the situation prior to treatment.
  5. Negative sensitivity recorded at recall visit despite positive pulp response at baseline, or severe pain is noted. Removal of restoration and immediate root canal treatment is required or the tooth must be extracted.
Time Frame: 36 Months
Population: This population incudes all subjects that completed their three year visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
Number analyzed (Participants) | 35 | 34 | 34
Number analyzed (Teeth) | 35 | 34 | 34
units on a scale | 1.04 (0.19) | 1.04 (0.09) | 1.07 (0.27)
Statistical Analysis 1: Comparison: Universal Composite vs Flowable Composite vs Bulk Fill Flowable Composite; Test type: Superiority; p = 0.424, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Baseline through 36 months
Description: This was a split person design where each Subject received all three treatments. Only one Subject died, unrelated to study treatment. This death is reported for each of the three arms and so the sum total column indicates three deaths but it is actually only one.
Arm/Group | Universal Composite | Flowable Composite | Bulk Fill Flowable Composite
All-Cause Mortality (participants affected / at risk) | 1/53 | 1/53 | 1/53
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/53 | 1/53
Other Adverse Events (participants affected / at risk) | 3/53 | 2/53 | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Universal Composite (N=53) | Flowable Composite (N=53) | Bulk Fill Flowable Composite (N=53)
death (General disorders) | 1 | 1 | 1 — Principal Investigator did not specify cause of death.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Universal Composite (N=53) | Flowable Composite (N=53) | Bulk Fill Flowable Composite (N=53)
Loss of retention (General disorders) | 1 (1) | 0 (0) | 0 (0) — Loss of restoration (debond)
Restoration fracture (General disorders) | 2 (2) | 2 (2) | 2 (2)
Pulpitis (General disorders) | 0 (0) | 0 (0) | 2 (2) — Pulpitis followed by endodontic therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT02889835/Prot_SAP_000.pdf